CLINICAL TRIAL: NCT05937113
Title: A Cross-over, Open-label, Randomized Study Evaluating the Safety and Immunogenicity of the Inactivated Rabies Vaccine RABIVAX-S on Healthy Vietnamese Volunteers With 3 Doses of Pre-exposure Prophylaxis
Brief Title: Safety and Immunogenicity of the Inactivated Rabies Vaccine RABIVAX-S Administered Intramuscularly and Intradermally
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vietnam Military Medical University (Other)
Collaborators: Vabiotech (Industry)
Responsible Party: Principal Investigator, Pham Ngoc Hung, Department of Epidemiology, Vietnam Military Medical University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: VX.2019.02
Record Dates: First submitted 2023-06-29; First posted 2023-07-10 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Rabies
Keywords: Rabies; rabies vaccine; RABIVAX-S
MeSH Terms: conditions — Rabies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Safety of a 3-dose regimen of RABIVAX-S in healthy participants aged 5 to 60 years (Experimental): RABIVAX-S is a pure, sterile inactivated rabies vaccine produced on vero cells. RABIVAX-S vaccine is lyophilized and is supplied with rehydration solution (1 vial containing 1 dose of lyophilized vaccine and 1 vial of rehydration solution).
  Interventions: Biological: RABIVAX-S
- immunogenicityof a 3-dose regimen of RABIVAX-S in subgroup of participants (Experimental): RABIVAX-S is a pure, sterile inactivated rabies vaccine produced on vero cells. RABIVAX-S vaccine is lyophilized and is supplied with rehydration solution (1 vial containing 1 dose of lyophilized vaccine and 1 vial of rehydration solution).
  Interventions: Biological: RABIVAX-S

INTERVENTIONS:
Biological: RABIVAX-S — 1 ml dose vaccine containing ≥ 2.5 IU of purified rabies antigen (Pitman-Moore rabies virus strain 3218; acclimatized and cultured on vero cells, inactivated with β propiolactone).
  Pre-exposure prophylaxis regimens for two groups
  * Intramuscular 1ml on days D0, D7 and D21+7
  * Intradermal injection 0.1 ml on days D0, D7 and D21+7 Blood samples were collected on days D0, D7 and D21 - 28

SUMMARY:
Randomized, open-label, prospective, before-and-after comparison study in the same group.

Subjects suitable for the study will be randomly assigned at a ratio of 1:1 (block 4) to use the study vaccine by one of two routes of administration: Intramuscular or Intramuscular. Previously-unvaccinated subjects receive three injections of vaccine on day 0, 7 and 21-28. The aim of the study is to evaluate the safety and immunogenicity of the inactivated rabies vaccine RABIVAX-S administered intramuscularly and intradermally according to a 3-dose regimen in healthy volunteers.

DETAILED DESCRIPTION:
1 ml dose vaccine containing ≥ 2.5 IU of purified rabies antigen (Pitman-Moore rabies virus strain 3218; acclimatized and cultured on vero cells, inactivated with β propiolactone).

Pre-exposure prophylaxis regimens for two groups

* Intramuscular 1ml on days D0, D7 and D21-28
* Intradermal injection 0.1 ml on days D0, D7 and D21-28

Randomization was performed according to two age stratifications:

* Stratification of research subjects from 5-15 years old
* Stratification of research subjects from 16-60 years old Population selected research subjects in the community in Dong Hung district, Thai Binh province

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers aged 5-60 years at the time of study screening.
2. Consent to participate in the study by signing the consent to participate in the study after being provided with complete information about the study. The participation of research subjects under the age of 18 years will be signed by the legal guardian.
3. Research subjects with normal health are determined according to personal medical history, clinical examination and laboratory tests within the clinically acceptable normal range.
4. Able to follow the research process as assessed by the researcher.
5. Women of reproductive age who have been using effective contraception for at least 4 weeks prior to screening and are willing to continue contraception until at least 4 weeks after the last dose of the study vaccine together. Men participating in the study agreed not to conceive until at least 4 weeks after the last dose of the study vaccine.

Exclusion Criteria:

1. Subject is participating in any other clinical trial.
2. Research facility staff working directly in this study and their families and relatives. Family, relatives are defined as spouses, parents, children or siblings, whether adopted or legally adopted.
3. History of previous rabies vaccination (pre- or post-exposure regimen)
4. Have received rabies immunoglobulin (human/equine) in the past.
5. Fever (temperature ≥37°C) or moderate or severe acute illness, or infection on the day of vaccination.
6. History of systemic hypersensitivity reaction to any vaccine component or history of life-threatening reaction to an experimental vaccine or a vaccine containing any vaccine-like substance study.
7. Have received any immunoglobulin, blood, or blood-based product therapy in the past 3 months, which may interfere with the assessment of immune response.
8. Known seropositive status for HIV antibody, HCV antibody or hepatitis B surface antigen (HBsAg) (retest not required).
9. Receive any vaccine in the 4 weeks before the first trial vaccine
10. Expect to receive any vaccine for 4 weeks after the trial vaccine is administered.
11. Women who are pregnant or have a positive urine test or are not willing to use safe methods of contraception
12. Women who are breastfeeding
13. Participated in a clinical trial study within the past 3 months.
14. Have a plan to donate blood while participating in the study
15. History of or current drug or alcohol abuse within the past year.
16. Congenital or acquired immunodeficiency, immunosuppressive therapy such as antineoplastic chemotherapy or radiation within the previous 6 months, or long-term systemic corticosteroid therapy (Permission to use topical steroid/medication)
17. Thrombocytopenia, bleeding disorders or anticoagulants in the 3 weeks prior to vaccination is contraindicated intramuscularly (IM)
18. Subjects at high risk of exposure to rabies during the study period, for example veterinary surgeons (including students at veterinary colleges), technical staff working with doctors veterinarians, laboratory staff handling rabies-contaminated material, abattoir staff, zoo staff.
19. Subject plans to have surgery in the next 3 months.
20. Subjects using antimalarial drugs concurrently
21. Clinically significant acute or chronic conditions such as pulmonary, endocrine, autoimmune, psychiatric, cardiovascular, liver or renal disease, as determined by medical history and physical examination and in the opinion of the researcher may affect the objectives of the study.
22. Any other condition that, in the opinion of the researcher as a member, would jeopardize the safety or rights of the subject or prevent the subject from completing the protocol procedures study.

Ages: 5 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 220 (Actual)
Dates: Start 2020-06-13 (Actual); Primary Completion 2020-07-02 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Rate of Subjects Experiencing Solicited Local and Systemic Adverse Events (AE) after | Within 30 minutes of each vaccination
  Solicited local and systemic AEs were assessed by study staff in 30 minutes after vaccination.
Rate of Subjects Experiencing Solicited Local and Systemic Adverse Events (AE) | within 7 days (day 1 to 7) of each vaccination and within 21 day after the first vaccination
  Solicited local AEs were assessed by study staff 30 minutes after vaccination then daily for 7 days
Rate of Subjects Experiencing Unsolicited Adverse Events (AE) | during 21 days after the third vaccination
  Unsolicited AEs were observed by study staff while the subject is at a clinic for a study visit or reported by the subject at any time. Any sign or symptom that would normally be considered a "solicited AE" (for example, fever, nausea, injection site pain) starting after 7 days post-vaccination was to be recorded as an unsolicited AE
Rate of Subjects Experiencing Unsolicited Serious Adverse Events (SAE) | Day 1 to Day 42
  A serious adverse event (SAE) is defined as an AE that meets one of the following conditions:
  Deadly. Life-threatening. Requires inpatient hospital admission or extended stay in hospital. Causes birth defects. Causes permanent or permanent injury or disability. Critical medical events that may not be fatal, not life-threatening, or require inpatient treatment will be considered a SAE if it is judged by professional judgment that the incident would be potentially dangerous. subject's health and the need for medical or surgical intervention to prevent one of the aforementioned consequences

SECONDARY OUTCOMES:
Rate of Subjects With Seroconversion of rabies virus neutralizing antibody (RVNA) for Vaccine Antigens for subgroup of subjects | Day 0, day 7, day 21 and day 42
  Serum specimens were tested for the presence and titer of rabies virus neutralizing antibody (RVNA) and the seroprotection rate was RVNA titer ≥0.5 IU/mL
Geometric Mean Titer (GMT) of rabies virus neutralizing antibody (RVNA) for Vaccine Antigens at Baseline and Day 22 or 49 after vaccination (depending on age group) for each antigenic component of the vaccine | Day 0, day 7, day 21 and day 42
  Serum specimens during Phase 3 were tested for the presence and titer of RVNA

CONTACTS AND LOCATIONS:
Overall Officials: Pham N Hung, As. Prof., Principal Investigator — Vietnam Military Medical University
Locations (1):
- CDC Thai Binh, Thái Bình, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hung PN, Giang LTH, Anh NT, Anh BDT, Pho DC, Van Hung P. Safety and immunogenicity of an inactivated vero cell-based rabies vaccine (Rabivax-S) in pre-exposure prophylaxis schedule in Vietnam. Clin Exp Vaccine Res. 2025 Jan;14(1):51-58. doi: 10.7774/cevr.2025.14.e9. Epub 2025 Jan 22. PMID 39927222